CLINICAL TRIAL: NCT04351867
Title: The Efficacy and Safety of Postoperative Chemotherapy With Docetaxel Plus Oxaliplatin and Capecitabine Versus Oxaliplatin Plus Capecitabine for Postoperative Pathological Stage IIIB/IIIC Gastric Adenocarcinoma: a Randomised, Phase 3 Trial
Brief Title: A Clinical Trial of Two Adjuvant Chemotherapy Regimens for Postoperative Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LiNing (Other Government)
Responsible Party: Sponsor-Investigator, LiNing, Chief Physician, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC202001
Record Dates: First submitted 2020-03-27; First posted 2020-04-17 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): docetaxel plus oxaliplatin and capecitabine
  Interventions: Drug: docetaxel plus oxaliplatin and capecitabine
- control group (Active Comparator): oxaliplatin plus capecitabine
  Interventions: Drug: oxaliplatin plus capecitabine

INTERVENTIONS:
Drug: docetaxel plus oxaliplatin and capecitabine — docetaxel 50mg/㎡ ivgtt. d1+oxaliplatin 100mg/㎡ ivgtt. d1+capecitabine 1000mg/㎡ bid p.o. d1-d14 q21d
  Other Names: Three medicine combined
  Arms: experimental group
Drug: oxaliplatin plus capecitabine — oxaliplatin 130mg/㎡ ivgtt. d1+capecitabine 1000mg/㎡ bid p.o. d1-d14 q21d
  Other Names: Two medicine combined
  Arms: control group

SUMMARY:
This study was a prospective, randomized, controlled phase III clinical study to evaluate the efficacy and safety of docetaxel plus oxaliplatin and capecitabine versus oxaliplatin plus capecitabine in the treatment of gastric or gastroesophageal junction adenocarcinoma with postoperative pathological stage IIIB and IIIC.

DETAILED DESCRIPTION:
In 2019, CSCO guidelines grade I recommend gastric or gastroesophageal junction adenocarcinoma patients, after D2 R0 resection, whose postoperative pathological stage was III treated with XELOX as an adjuvant chemotherapy. However, some retrospective clinical studies in China suggest that the 3-year DFS rate of XELOX program as an adjuvant postoperative chemotherapy program is still low, and the risk of recurrence is higher for patients with postoperative pathological stage IIIB/IIIC.In recent years, the success of the JACCRO GC-07 trial has provided evidence for the value of Taxoids in postoperative adjuvant therapy of gastric cancer. In the FLOT4 trial, the FLOT improved the DFS rate by 3 years compared with the ECF/ECX. At present, there is no clinical study data to prove whether the combined three-drug regimen can further reduce the risk of postoperative recurrence and improve the treatment effect compared with oxaliplatin combined capecitabine two-drug regimen for patients with high postoperative recurrence risk (patients with postoperative pathological stage IIIB/IIIC). Therefore, the investigators carried out this trial.

ELIGIBILITY:
Inclusion Criteria:

* Have signed the informed consent and can comply with the visit and related procedures stipulated in the program
* Age ≥18 years old and ≤75 years old
* D2 radical resection was performed within 21-60 days before the beginning of the first cycle of chemotherapy in this clinical study
* Preoperative neoadjuvant chemotherapy was not performed and Gastric and gastroesophageal junction adenocarcinoma (including signed-ring cell carcinoma, mucinous adenocarcinoma, and hepatoid adenocarcinoma) at stage IIIB and IIIC were confirmed by postoperative pathological staging. Note: the presence of distant metastases should be confirmed by a CT or MRI scan.ECT should be performed if bone metastases are suspected.If peritoneal metastases are suspected, laparoscopy should be performed
* Postoperative ECOG score was 0 or 1
* Leukocyte ≥ 4×109/L, platelet ≥ 100×109/L without blood transfusion, neutrophil absolute value (ANC) ≥ 1.5×109/L without granulocyte stimulating factor treatment, and hemoglobin ≥ 90 g/L
* Bilirubin ≤ 1.5 times of the upper limit of normal value, glutamic oxalacetic transaminase and glutamic-pyruvic transaminase ≤ 2.5 times of the upper limit of normal value
* Serum creatinine ≤ 1.5 times the upper limit of normal value, or GFR>45 ml/min
* Serum albumin ≥ 25 g/L (2.5g /dL)
* INR or PT ≤ 1.5 times ULN
* Hepatitis b surface antigen positive patients need to be tested for hepatitis b DNA virus quantitative detection, only < the upper limit of the normal detection value can be included in the group, and should long-term use of anti-hepatitis b drugs
* Tumor specimens can be provided for consultation (if the patient's surgical specimen comes from another hospital), protein and gene testing

Exclusion Criteria:

* Postoperative wound healing is poor and chemotherapy is not appropriate to start
* Recurrent patients or suspected peritoneal metastases after radical surgery
* Known DPD enzyme deficiency
* Allergy to, or history of severe allergy to, or contraindication to any of the experimental drugs or its excipients
* Patients who are expected to require major surgery during the study period
* Congenital pulmonary fibrosis, drug-induced pneumonia, organized pneumonia, or CT-confirmed active pneumonia
* Tested positive for HIV
* Active hepatitis b or c
* Only liquid diet was allowed after the operation, with BMI <18kg/m2
* Uncontrolled pain
* A history of antitumor drug therapy other than radical surgery
* Severe infection in the active stage or with poor clinical control
* Use of hormones is contraindicated
* Severe cardiovascular disease, myocardial infection or cerebrovascular accident, arrhythmia, unstable angina pectoris within 3 months before the trial
* Uncontrollable increase in blood pressure or blood sugar
* A history of other malignancies within 5 years, except for carcinoma in situ of the cervix, non-melanoma skin cancer, or stage I uterine cancer
* Distant metastases are known
* Peripheral neuropathy ≥ NCI CTCAE grade 2
* Serum albumin < 2.5 g/dL
* Chronic enteritis
* Any other disease for which there is evidence of a need to limit the use of experimental drugs
* Participate in additional trials up to 30 days before the trial or plan to participate in additional trials while the trial is ongoing
* Receive other experimental drugs up to 28 days before the start of the trial
* Women who are pregnant or nursing, or who plan to become pregnant within five months of the end of treatment. Women of childbearing age should receive a blood/urine pregnancy test 7 days before the start of the trial
* Clinically significant active bleeding
* Patients who have trouble swallowing tablets
* Previous allogeneic bone marrow transplant or organ transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
disease free survival | up to three years.
  From the date of randomization until the date of the first recorded disease recurrence, metastasis or death from any cause, whichever came first.

SECONDARY OUTCOMES:
overall survival | up to three years.
  From the date of randomization until the date of the first recorded death from any cause. For subjects lost to follow-up prior to death, the last follow-up time is usually calculated as the time of death.
Adverse reaction | up to three years.
  Adverse reaction will be assessed by NCI CT CAE v5.0.
Assessment of life quality | up to three years.
  Quality of life will be assessed using The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Cancer (QLQ-C30) and the site-specific module for gastric cancer (QLQ-STO22) . These tables will be usde together to assessed the quality of life of the patients. The higher the score, the worse the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, PhD, Principal Investigator — Henan Cancer Hospital; Suxia Luo, PhD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Raw data
Time Frame: Within 1 year after completion of the main part
Access Criteria: public management platform ResMan (www.medresman.org) was adopted to provide open access to the public